CLINICAL TRIAL: NCT04839705
Title: Post-Approval Study - Post-Market Surveillance Study to Evaluate the Long-Term Safety and Effectiveness of the WEB Device
Brief Title: Post Approval Study - Evaluate the Long-Term Safety and Effectiveness of the WEB Device
Acronym: WEB PAS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Microvention-Terumo, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CL11010-001
Record Dates: First submitted 2021-04-07; First posted 2021-04-09 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Wide Neck Bifurcation Intracranial Aneurysms
Keywords: Aneurysm; Intracranial Arterial Disease; Cerebrovascular Disorders
MeSH Terms: conditions — Aneurysm; Intracranial Arterial Diseases; Cerebrovascular Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- WEB Aneurysm Embolization Device (Other): WEB Aneurysm Embolization Device The WEB is an intra-aneurysmal device intended for use in endovascular embolization of intracranial aneurysms. The intended therapeutic effect of the WEB device is to line the neck of the aneurysm with a metallic structure that disrupts the inflow of blood, causing hemostasis within the aneurysm sac, and leading to thrombus formation within the implant.
  Interventions: Device: WEB

INTERVENTIONS:
Device: WEB — Device: WEB The WEB is an intra-aneurysmal device intended for use in endovascular embolization of intracranial aneurysms.
  Other Names:
  • WEB Aneurysm Embolization Device

SUMMARY:
A prospective, multicenter, single arm, interventional study. The target patient population for this study are adult subjects with WNBAs of the anterior and posterior intracranial circulation. The primary effectiveness outcome of the study is adequate intracranial aneurysm occlusion on the 1 year angiogram as adjudicated by a core laboratory.

ELIGIBILITY:
Key Inclusion Criteria:

* Patient must be ≥ 18 at the time of screening
* Patient must have a single ruptured or unruptured IA requiring treatment
* Patient must sign and date an IRN approved written informed consent prior to initiation of any study procedures

Key Exclusion Criteria:

* Patient has an IA with characteristics unsuitable for endovascular treatment
* Patient has conditions placing them at high risk for ischemic stroke or has exhibited ischemic symptoms such as transient ischemic attacks, minor strokes, or stroke-in-evolution within the prior 30 days
* Patient has had an SAH from a non-index IA or other intracranial hemorrhage within 90 days
* Patient index IA was previously treated
* Patient is pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2022-08-24 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Key Effectiveness Outcome | 12 Months
  Proportion of subjects with adequate aneurysm occlusion at one year after treatment.
Key Safety Outcome | 12 Months
  Proportion of subjects with death of any nonaccidental cause or any major stroke* within the first 30 days after treatment or major ipsilateral stroke or death due to neurologic cause from day 31 to the 1 year after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Adam Arthur, MD, Principal Investigator — Methodist University Hospital, Memphis TN; David Fiorella, MD, Principal Investigator — Stony Brook University, Stony Brook NY
Locations (29):
- United States (29):
  - Memorial Health Systems, Hollywood, Florida
  - Orlando Health Neuroscience Institute, Orlando, Florida
  - The Queen's Medical Center Neuroscience Institute, Honolulu, Hawaii
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Kansas Health System, Kansas City, Kansas
  - Baptist Health Systems, Lexington, Kentucky
  - University of Kentucky, Department of Neurosurgery, Lexington, Kentucky
  - Norton Healthcare, Louisville, Kentucky
  - LSU Health Sciences Center at Shreveport, Shreveport, Louisiana
  - University of Maryland, Baltimore, Baltimore, Maryland
  - Johns Hopkins University, Baltimore, Maryland
  - Massachusetts General Brigham Incorporated, Boston, Massachusetts
  - UMass Memorial Health, Worcester, Massachusetts
  - Abbott Northwestern Hospital Allina Health, Minneapolis, Minnesota
  - The Washington University, St Louis, Missouri
  - Albany Medical Center, Albany, New York
  - University of Buffalo, Buffalo, New York
  - Northshore University Hospital/Northwell Health, Manhasset, New York
  - SUNY Stony Brook, Stony Brook, New York
  - Montefiore Medical Center, The Bronx, New York
  - Duke University, Durham, North Carolina
  - Ohio State University, Columbus, Ohio
  - OhioHealth Research Institute, Columbus, Ohio
  - The Toledo Hospital d/b/a ProMedica Toledo Hospital, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - University of Pennsylvania Health Systems, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Semmes Murphey, Memphis, Tennessee
  - West Virginia University, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: No